CLINICAL TRIAL: NCT06929143
Title: Real-world Utilization Patterns of Aflibercept 8 mg in Japan: a Retrospective Descriptive Study Using the Claims Database
Brief Title: A Study to Learn More About the Use of Aflibercept in Routine Medical Practice in Japanese Participants With Neovascular Age-related Macular Degeneration and Diabetic Macular Edema
Status: Active, not recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22905
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Neovascular Age-related Macular Degeneration (nAMD); Diabetic Macular Edema (DME)
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with neovascular Age-related Macular Degeneration (nAMD): Patients with any International Classification of Diseases, Tenth revision (ICD-10) codes for nAMD or possible nAMD within the same month of the cohort entry date (except for patients who meet the nAMD/DME cohort definition).
  Interventions: Drug: Aflibercept (Eylea, BAY86-5321)
- Patients with Diabetic Macular Edema (DME): Patients with any ICD-10 codes for DME or possible DME within the same month of the cohort entry date (except for patients who meet the nAMD/DME cohort definition).
  Interventions: Drug: Aflibercept (Eylea, BAY86-5321)
- Patients with nAMD/DME: Patients who have ICD-10 codes for nAMD, possible nAMD, DME, and possible DME within the same month of the cohort entry date.
  Interventions: Drug: Aflibercept (Eylea, BAY86-5321)
- Other patients: Patients with no ICD-10 codes for nAMD, possible nAMD, DME, and possible DME within the same month of the cohort entry date.
  Interventions: Drug: Aflibercept (Eylea, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept (Eylea, BAY86-5321) — 8 mg (0.07 mL) intravitreal (IVT) injection (114.3mg/mL).

SUMMARY:
This is an observational study in which data already collected from participants with neovascular age-related macular degeneration (nAMD) or diabetic macular edema (DME) is studied. In observational studies, only observations are made without participants receiving any advice or any changes to healthcare.

The eye disorders, nAMD and DME, affect the macula, the central part of the retina at the back of the eye. This leads to blurry vision or blind spots, making everyday activities like reading or sewing difficult. While nAMD is linked to aging, DME is related to diabetes. Both conditions require similar treatment to help improve vision.

Aflibercept 8 milligrams (mg) is already approved in Japan for doctors to prescribe to people with nAMD or DME. It is a drug injected into the eye. It works by blocking a protein called vascular endothelial growth factor (VEGF), which causes abnormal growth and leakage of blood vessels at the back of the eye.

The participants in this study are already receiving treatment with aflibercept 8 mg as part of their regular care from their doctors.

There is limited data available on the use of aflibercept 8 mg in Japan. Data from routine medical practice will inform treatment in Japanese and other Asian populations.

The main purpose of this study is to learn more about the disease and patient characteristics of Japanese participants with nAMD and/or DME who receive aflibercept 8 mg during their routine healthcare, and how they use it.

To learn this, the study will use 2 methods:

Method 1: Researchers will study the health details of participants when they first started aflibercept 8 mg.

Method 2: Researchers will study the participants' data collected over 1 year to see how they used aflibercept 8 mg.

The data will come from a claims database called DeSC Healthcare Inc. The data will be collected from April 2023 to March 2025 for Method 1, and from April 2023 to March 2026 for Method 2.

Researchers will only look at the information from participants in Japan.

In this study, only available data from routine care are collected. No visits or tests are required as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are prescribed aflibercept 8 mg during the observable period from the collected data.

Exclusion Criteria:

* Patients in the nAMD cohort or nAMD and DME cohort who have the ICD-10 codes for nAMD who are aged <40 years old.
* Patients in the DME cohort or others who are aged <18 years old.
* Female patients who have any pregnancy-related records.
* Patients who do not have at least 365 days of continuous enrollment in the database.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples will be taken from the DeSC healthcare insurance database. This database contains information of 12 million individuals and has in a previous study been found to be demographically distributed in a similar manner to the Japanese population.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Description of baseline characteristics of patients with nAMD or DME who initiated aflibercept 8 mg under real-world conditions. | At baseline.
Description of the longitudinal patterns of treatment interval of patients with nAMD or DME who initiated aflibercept 8 mg. | Within 12 months.

SECONDARY OUTCOMES:
Change of treatment interval of patients with nAMD or DME who are treated with other anti-VEGF therapy. | Before and 12 months after initiation of aflibercept 8 mg.
Number of injections of aflibercept 8 mg in patients with nAMD or DME. | Within 3 months, 6 months, and 12 months after the first prescription date of aflibercept 8 mg.
Predicting factors of the patterns of the treatment interval of aflibercept 8 mg in patients with nAMD or DME. | Within 12 months.
Proportion of patients who continue the aflibercept 8 mg. | Within 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Bayer, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.